CLINICAL TRIAL: NCT03117582
Title: Fecal Microbiota Transplantation (FMT) in Clostridium Difficile Infection (CDI) Not Responding to Antibiotics
Acronym: FMT
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other); North Carolina State University (Other)
Responsible Party: Sponsor
Other Study IDs: 16-2283
Record Dates: First submitted 2017-03-11; First posted 2017-04-18 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Clostridium Difficile
Keywords: C. diff; CDI; Clostridium Difficile Infection; Diarrhea; Fecal microbiota transplantation; FMT
MeSH Terms: conditions — Clostridium Infections; Diarrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — donor stool (25mL aliquot) stool specimen (4 samples, each ~3mL)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with C.diff infection: Patients with C.diff infection not responding to antibiotics who are now scheduled for the FMT procedure for routine care of their condition.
  Interventions: Other: Stool specimen

INTERVENTIONS:
Other: Stool specimen — The following stool specimen will be collected for this study:
  1. 4, 3mL stool specimen from patient
  2. 1, 25mL stool aliquot from donor

SUMMARY:
Purpose: To study the changes in the microbiome and stool composition in patients with Clostridium Difficile Infection (CDI) who undergo Fecal Microbiota Transplantation (FMT), along with changes in their clinical characteristics.

DETAILED DESCRIPTION:
This is a prospective, descriptive cohort study. Patients will receive current standard of care.

Once a potential subject is planned for FMT, they will be approached by study coordinators or investigators for participation in the study. If they agree to participate in the study, then patient health, medical and demographic information will be collected from the patient and/or from the medical record and entered into the research database, and associated with a research code with which the stool samples will also be labeled.

The study coordinator will be responsible for ensuring completion of the study questionnaire, which consists of pre- and post-FMT sections. The questionnaire will be attempted to be administered in person by the physician or study coordinator at a clinic visit, but may on occasion be completed at home and mailed in to the study coordinator or physician, or completed over the phone with the study coordinator or physician.

Stool preparations will be obtained by a nonprofit third party, OpenBiome, with whom the University of North Carolina has collaborated for over one year. Preparations include a 250mL (milliliter) preparation for lower administration, a 30mL preparation for upper administration, and frozen capsules (30 in one treatment) for oral delivery.

The actual FMT procedure will be performed in the majority of cases by colonoscopy. Other possible routes of administration are via nasogastric or nasoduodenal tube (with upper formulation), enema and frozen oral tablets. The current preferred route of administration is via colonoscopy, based on observation (no head-to-head) trials showing improved efficacy, but standards of care may change in the future. In all cases, the route of administration will be based on patient characteristics and preferences, not for purposes related to the study. In all cases, informed consent for the treatment will be documented as guided by the Food and Drug Administration (FDA). The patient will stop all antibiotics (including vancomycin or other antibiotics against C. diff) at least 2 days prior to FMT. For all administrations other than oral capsules, patients will perform a bowel preparation with 4 liters of Golytely or equivalent osmotic laxative split between the evening prior to the procedure and the morning of the procedure. In a minority of instances, especially for pediatric patients, the patient may be electively admitted to the hospital the night before, to monitor medical stability during the preparation, facilitate bowel preparation, and provide intravenous hydration. The bowel cleansing preparation is generally taken orally, though in rare instances must be administered via nasogastric or nasoduodenal (NG/ND) tube. Hospital admission and bowel preparation via NG/ND tube will only be performed if indicated as standard-of-care, not for purposes specifically related to the study.

For colonoscopic FMT, the procedure will be performed with anesthesia support at the UNC Memorial Hospital endoscopy unit. Sedation will be at the discretion of the treating anesthesiologist in agreement with the endoscopist, but generally consists of intravenous propofol, with monitored anesthesia care. For colonoscopic FMT, the patient is given two 2mg doses of loperamide orally, two hours prior to FMT, and is then to take an additional two capsules after recovery from anesthesia (recommended immediately upon arrival home, when an outpatient procedure).

Donor stool is obtained from OpenBiome, a third-party stool bank that screens donors for medication use, allergies, and health-related conditions and prepares stool per a standard protocol including suspension in normal saline. 250ml of donor stool is used for colonoscopic FMT in patients with over one meter squared of body surface area. For small children this quantity may be reduced proportionately. The entire 250ml's are placed into the ileum, cecum and/or ascending colon, or at the extent reached by the colonoscope, via the operative channel of the colonoscope. Patients are asked to maintain a right lateral recumbent position as much as possible for the hour after infusion, to encourage permanence of the material in the proximal colon. Of note, the FMT colonoscopy does not include meticulous mucosal examination if not otherwise indicated, and as such is not a substitute for routine colorectal cancer screening. Patients are monitored by post-anesthesia care unit (PACU) personnel until ready for discharge, per standard unit protocol.

For nasogastric or nasoduodenal administration, 30ml of donor stool is infused slowly over 1 hour. Before infusion, NG/ND tube placement is confirmed by X-ray per standard hospital protocol, according to standard hospital consent form.

In rare cases where procedural sedation, colonoscopy or NG/ND tube is contraindicated, frozen oral capsules or enema may be used to administer FMT. With capsule administration, in addition to stopping antibiotics two days prior to the procedure, the patient takes proton pump inhibitor on the day before treatment and the day of treatment. There is no bowel preparation. The patient takes the 30 capsules orally under direct physician supervision within 90 minutes. Metoclopramide 5-10 mg x i may be taken one hour prior to the treatment. With enema administration, bowel preparation will be performed prior to administration. Bowel cleansing preparation, loperamide administration, and right lateral recumbency will be attempted as per colonoscopic FMT. The enema will be administered under direct physician supervision, as well.

For the study, subjects who are undergoing the above treatment per standard of care will be asked to submit four (4) total stool samples. The first will be pre-FMT, at any time from 2 weeks prior to FMT (possibly at a clinic visit), up until directly before the pre-FMT bowel preparation. Post-FMT stool samples at 2 weeks (range 1-3 weeks), 2 months (range 7-9 weeks) and 6 months post-FMT.

All stool samples will be collected according to the same protocol, described in a handout (entitled "Stool Collection Instructions") provided to participants. There are several options for submitting the sample, basically according to patient convenience. If they can produce a sample at a clinic visit, they can submit at that time. Alternatively, they will be provided supplies to safely collect and then store samples they collect at home in their own freezer. They will then have to deliver these samples to UNC (or possibly North Carolina State University [(NCSU)] if that is more convenient for a particular subject), which can be done at one visit with all of the samples, or in segments as they collect them. Before submission to the biobank, the samples will be labeled with the research code and any other identifying labels on the stool sample will be removed and destroyed. The de-identified stool specimens will be aliquoted in the research laboratory for storage at -80° Celsius.

They will be transported by the study coordinators from UNC to a storage unit at NCSU. Research samples will be stored in a manner that will permit subsequent microbial DNA extraction, microbial cultivation and metabolite analysis.

They will also be asked to complete a post-FMT section of the questionnaire, from which the main outcomes of FMT will be determined. They will be evaluated at two post-FMT clinic visits, which may correspond to first two post-FMT stool samples, where evidence for any possible adverse events or recurrences will be personally queried and evaluated. If patients do not attend any scheduled post-FMT visits, the study coordinator will attempt to contact them by phone and then by mail, both to encourage them to reschedule their clinic visit, of if this is not possible, then to at least obtain the questionnaire data.

Primary aim (clinical outcomes): Descriptive statistics of the clinical outcomes, such as mean and median number of days of symptom duration, primary cure rate, percentage of subjects with resolution of diarrhea, abdominal pain, fatigue, etc will be calculated. Standard deviations and/or confidence intervals will be provided where appropriate. If statistical power allows, multivariate logistic regression models may be used to identify patient-level risk factors predictive of primary cure (such as sex, age, independent-living status, etc.).

Secondary aims: Differences in pre-and post-FMT stool composition, and between early and late post-FMT samples, will be calculated with McNemar's test for significant differences in proportions of rRNA (ribosomal ribonucleic acid) sequences pertaining to the relevant bacterial phyla (Bacteroidetes, Firmicutes, and Proteobacteria), and paired t-tests and ANOVA's (or their non-parametric counterparts) for significant differences in Shannon diversity indices (a measure of bacterial diversity) and in concentrations of multiple bile acids. If these measures are different from pre- to post-FMT samples, then the relationship of percent differences in each stool parameter to clinical outcome will be evaluated using logistic regression with primary outcome of "primary cure" within two months of FMT, and a Cox proportional hazards model with the time variable as "days to primary cure" and the censor variable as "primary cure." Secondary analyses may be conducted with "any cure" as the outcome variable if repeat FMT is frequently needed. The investigators will also compare a sample of donor stool to the post-FMT samples with the same statistical tests, under the hypothesis that the closer that post-FMT stool resembles donor stool (and the more durable this resemblance), the better the clinical response. All statistical analyses will be performed at an alpha of 0.05.

ELIGIBILITY:
Inclusion criteria:

1. As subjects must meet standard clinical criteria for candidacy for FMT, all patients will have suffered symptomatic diarrhea and have documented stool c. difficile toxin positivity. Almost all patients will have failed standard therapy for CDI, which includes at least one course of treatment with a primary agent (metronidazole, vancomycin or fidaxomicin), as well as an extended vancomycin taper following either the second or third recurrence. There may be extenuating circumstances that could justify FMT for CDI outside of these parameters, such as severe allergy to multiple of the above agents, though this would be expected to be exceedingly rare.
2. All patients must be able to tolerate either colonoscopy (including anesthesia and sedation) or placement of a nasogastric/nasoduodenal tube, without a contraindication to the procedure.

Exclusion criteria:

1. Pregnancy
2. Prisoners (for concerns of vulnerability and logistics)
3. Adult patients who are themselves unconsentable at time of FMT.
4. Life expectancy judged to be <3 months
5. Need for extended antibiotics at baseline, for an indication other than treatment for CDI
6. Any patient who the clinician judges to be a poor candidate for FMT, for reasons of comorbidities or not being able to tolerate the procedure for administration, would by definition be excluded from the study.

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are receiving FMT procedure at UNCH and meet the eligibility criteria below:
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-05-02 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
Percent of participants who had resolution of diarrhea. | 8 weeks after FMT procedure
  Diarrhea is defined as three or more unformed stools for more than two consecutive days.

SECONDARY OUTCOMES:
Percent of participants who did not need antibiotics to treat diarrhea. | 8 weeks after FMT procedure
  Antibiotic use for C. difficile infection after the FMT procedure will be documented.
Difference in stool microbiome before and after FMT procedure. | 6 months after FMT procedure
  Difference is defined as the proportion of bacterial rRNA sequences belonging to the phyla 1) Bacteroidetes, 2) Firmicutes, and 3) Proteobacteria at pre-treatment, two weeks post, 2 months post, and 6 months post FMT procedure.
Difference in stool metabolome before and after FMT procedure. | 6 months after FMT procedure
  Difference is defined as the concentration of bile acids (cholic, lithocholic, deoxycholic, chenodeoxycholic, taurocholic and taurochenodeoxycholic acids) in mg/g at pre-treatment, two weeks post, 2 months post, and 6 months post.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay S Gulati, MD, Principal Investigator — UNC Chapel Hill
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States